CLINICAL TRIAL: NCT06679205
Title: Effectiveness of a Multidisciplinary Treatment for Patients With Chronic Low Back Pain (PAINDOC Protocol): Randomized, Parallel-group, Two-arm, Single-blind Clinical Trial (PAINDOC Project)
Brief Title: Effectiveness of a Multidisciplinary Treatment for Patients With Chronic Low Back Pain
Acronym: PAINDOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Anna Dalmau Roig, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2024/0791
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low-back Pain (cLBP); Chronic Low-back Pain; Back Pain
Keywords: chronic low-back pain; chronic pain; pain catastrophizing; multidisciplinary treatment; therapeutic exercice; pain neuroscience education; cognitive behavioural therapy; therapeutic education
MeSH Terms: conditions — Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacological control (Active Comparator): The subjects in the control group will be treated following a pharmacological approach according to the latest clinical guidelines for patients with chronic low back pain. Thus, the pharmacological options to be considered in each patient will be those included in the first and second analgesic steps of the WHO (preferably without including minor opioids).
  Interventions: Drug: Usual Care
- PAINDOC program (Experimental): The PAINDOC Program is a multidisciplinary treatment that integrates four parts provided by different health professionals and consists of 7 sessions carried out in the pain unit of the Hospital Clinic of Barcelona over 2 months. It consists of a therapeutic education session (Empowered Relief®) given by a physician from the unit, a pain psychology session given by a psychologist, and 2 pain neuroscience education sessions and 3 therapeutic exercise sessions given by a physiotherapist. This program is already part of the pain unit's routine care practice, so it is considered that the sessions of this program do not represent an additional and specific visit for the patients.
  Interventions: Behavioral: Multidisciplinary and multimodal intervention

INTERVENTIONS:
Behavioral: Multidisciplinary and multimodal intervention — The PAINDOC Program consists in:
  * Therapeutic education: The therapeutic education block consists of 2 parts: a 2-hour education session called Empowered Relief® and 2 1-hour pain neuroscience education sessions.
  * Psychotherapy: The psychotherapy part consists of 1 group session of 1 hour, face-to-face and with groups of up to 15 people.
  * Therapeutic exercise: The therapeutic exercise module consists of 3 sessions of 1 hour each, face-to-face, with small groups of between 6 and 10 patients, and given by the physiotherapist of the pain unit.
  Other Names: PAINDOC program
  Arms: PAINDOC program
Drug: Usual Care — The pharmacological treatment will be individualised according to pain intensity, contraindications and the appearance of adverse effects.
  Other Names: Pharmacological Control
  Arms: Pharmacological control

SUMMARY:
PAINDOC is a treatment program that includes 4 disciplines that, separately, have demonstrated their effectiveness in the treatment of chronic low back pain: education in pain neuroscience, therapeutic education (Empowered Relief®), psychotherapy based on cognitive-behavioral therapy and therapeutic exercise.

The primary objective of the study is to evaluate the effectiveness of the PAINDOC multidisciplinary treatment program in reducing pain intensity and improving quality of life in persons with chronic low back pain referred to the pain unit of the Hospital Clinic of Barcelona, compared to usual care treatment.

As secondary objectives, the present study aims to evaluate the effect of the PAINDOC program on:

* The reduction of pain-related disability.
* The reduction of pain catastrophizing.
* The improvement in perceived social support.
* The improvement in perceived autonomy (self-efficacy).
* The reduction of analgesic, anti-inflammatory and adjuvant analgesic medication.

The main questions it aims to answer are:

* Is the proposed multidisciplinary treatment effective in improving pain-related outcomes?
* Is the proposed multidisciplinary treatment effective in reducing analgesic medication?

Participants will receive either usual care (pharmacological control) or the PAINDOC program, which consists of 7 multidisciplinary sessions within 2 months. There will be one therapeutic education session called Empowered Relief®, 2 pain neuroscience education sessions, one pain psychology session and 3 therapeutic education sessions. Besides, participants will be assessed using written questionnaires before treatment, at 3 months and at 6 months.

Researchers will assess the effectiveness of the multidisciplinary treatment group comparing both groups to see if there is any difference in several pain-related outcomes.

DETAILED DESCRIPTION:
Despite improving pharmacological and surgical medical treatment options, chronic low back pain is the most frequent pain disorder and a leading cause of disability. Over the past decades, clinicians have acknowledged that a broader view of disease and disability is needed in chronic conditions treatment. Therefore, biological, psychological and social factors must be addressed to improve such conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with primary chronic low back pain (non-specific chronic low back pain) of axial predominance.
* Experiencing pain at least 50% of the time over the last 6 months.
* Average weekly pain intensity equal or greater than 4 out of 10 on a verbal numerical scale.
* Be agreeable to receiving active, non-pharmacological and non-surgical treatment.

Exclusion Criteria:

* Inflammatory low back pain.
* History of cancer in the last 5 years.
* Unexplained and unintentional weight loss of 10 Kg or more over the preceding 12-month period.
* Lack of control of bowel and bladder function (cauda equina).
* Difficulty in performing the sessions due to severe physical disability.
* Diagnosis of severe mental illness (schizophrenia, major depression, bipolar disorder, etc.).
* Strong prescription opioid or parenteral medication addiction disorders.
* Technical-logistical problems (inability to attend treatment sessions or inability to fill out assessment questionnaires).
* Problems in understanding the content of the sessions (language barrier, severe hearing loss or severe cognitive impairment).
* Have sought compensation or entered into litigation in the preceding 12-month period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity. Changes from baseline to 6 months. | Baseline, 3 months, 6 months
  Participants will be asked to rate their pain intensity on a horizontal 100-mm Visual Analogue Scale (VAS), ranging from 0 = no pain to 100 = worst imaginable pain. The VAS is a valid and reliable instrument compared with other pain rating scales, and has been well established in clinical practice and research for measuring pain levels in low back pain patients. For patients with subacute or chronic low back pain, the minimum clinically relevant change is considered to be at least 20 mm on a VAS.
Health-related quality of life. Changes from baseline to 6 months. | Baseline, 3 months, 6 months
  The spanish version of the Euro Quality of Life 5D-5L (EQ-5D-5L) was used to assess the health related quality of life (HRQL).(10) The EQ-5D-5L consists in two pages: the first one is based on a descriptive system that defines health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories: no problems, slight problems, moderate problems, severe problems, extreme problems.(10) A health state is composed by taking one level for each dimension, and a preference-based scoring function is used to convert the descriptive system to a summary index score (ranging from states worse than dead <0 to full health 1).

SECONDARY OUTCOMES:
Pain-related Disability. Changes from baseline to 6 months. | Baseline, 3 months, 6 months
  Disability will be assessed using the spanish version of the Oswestry Disability Index (ODI) questionnaire. The ODI is one of the most common specific measurement tools to evaluate the function and disability of lumbar spine pathologies. This questionnaire contains 10 items evaluated from 0 to 5 (higher values indicate greater disability), which correspond to 10 domains. The sum of the 10 scores is expressed as a percentage (ODI score), with ranges from 0% (no disability) to 100% (maximum disability).
Pain Catastrophizing. Changes from baseline to 6 months. | Baseline, 3 months, 6 months
  The Spanish version of Pain Catastrophizing Scale (PCS) was used to asses thoughts and feelings related to pain experiences.(9) The PCS is a 13 item self-administered questionnaire composed of 3 subscales: rumination, magnification and helplessness. The PCS uses a 5-point Likert scale with responses ranging from 0 = not at all to 4 = all the time. Overall scores range from 0 to 52 points, the higher the score, the higher is the pain catastrophism level.
Perceived Social Support. Changes from baseline to 6 months. | Baseline, 3 months, 6 months
  It will be assessed using the Lubben Social Network Scale (LSNS-6), which was developed to assess the perceived social support of an adult person according to the size of his or her social network, the trust that these ties generate and the frequency of contacts that this person has with those around him or her. The LSNS-6 includes 6 questions divided into 2 domains: 3 on family and 3 on friendships. It is one of the most widely used by the international community and its application is simple and brief, which is of vital importance for its feasibility in the clinical setting. The Spanish version of the LSNS-6 has proven to be valid and reliable.
Self-efficacy. Changes from baseline to 6 months. | Baseline, 3 months, 6 months
  Self-efficacy will be assessed using the Spanish version of the Chronic Pain Self-Efficacy Scale (CPSES). The CPSES is a 19-item self-administered questionnaire. Each item assesses the ability that the person believes he or she has to perform a certain task or activity and is presented in the form of a question. The person must consider each question on a 10-point Likert scale, with a range of 0 to 10, where 0 is "I think I am totally incapable" and 10 is "I think I am totally capable." The total score can range from 0 to 190 points, indicating greater self-efficacy in chronic pain the higher the score. This questionnaire is divided into 3 dimensions: self-efficacy in symptom control, self-efficacy in physical functioning, and self-efficacy in pain management.
Consumption of analgesic, anti-inflammatory and coadjuvant analgesic drugs | Baseline, 3 months, 6 months
  The doses of analgesic, anti-inflammatory and coadjuvant analgesic drugs taken by each participant will be recorded, expressed in mg/day, except for opioids, where the Morphine Equivalent Dose (MED) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Terradas-Monllor, PhD, Study Director — University of Vic; Christian Dürsteler, PhD, Study Director — University of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Bodes Pardo G, Lluch Girbes E, Roussel NA, Gallego Izquierdo T, Jimenez Penick V, Pecos Martin D. Pain Neurophysiology Education and Therapeutic Exercise for Patients With Chronic Low Back Pain: A Single-Blind Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):338-347. doi: 10.1016/j.apmr.2017.10.016. Epub 2017 Nov 11. PMID 29138049
- [Background] Vlaeyen JWS, Maher CG, Wiech K, Van Zundert J, Meloto CB, Diatchenko L, Battie MC, Goossens M, Koes B, Linton SJ. Low back pain. Nat Rev Dis Primers. 2018 Dec 13;4(1):52. doi: 10.1038/s41572-018-0052-1. PMID 30546064
- [Background] Darnall BD, Roy A, Chen AL, Ziadni MS, Keane RT, You DS, Slater K, Poupore-King H, Mackey I, Kao MC, Cook KF, Lorig K, Zhang D, Hong J, Tian L, Mackey SC. Comparison of a Single-Session Pain Management Skills Intervention With a Single-Session Health Education Intervention and 8 Sessions of Cognitive Behavioral Therapy in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2113401. doi: 10.1001/jamanetworkopen.2021.13401. Erratum In: JAMA Netw Open. 2022 Apr 1;5(4):e229739. doi: 10.1001/jamanetworkopen.2022.9739. PMID 34398206
- [Background] Ochandorena-Acha M, Dalmau-Roig A, Dursteler C, Vilchez-Oya F, Ferrer A, Martin-Villalba I, Obach A, Terradas-Monllor M. Acceptability of multimodal and multidisciplinary group-based program for chronic low back pain: a qualitative study. Physiother Theory Pract. 2025 May;41(5):981-997. doi: 10.1080/09593985.2024.2377343. Epub 2024 Jul 12. PMID 38994708
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143